CLINICAL TRIAL: NCT07238478
Title: Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy of JDS-HF3.0 in Menopause Related Quality of Life Outcomes in Postmenopausal Women
Brief Title: JDS-HF3.0 Supplementation on Menopause Related Quality of Life Outcomes in Postmenopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bonafide Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BH-TJP-BT-001; 13364-TAVanDusseldorp (Other: Sterling IRB)
Record Dates: First submitted 2025-05-06; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Joint Discomfort; Joint Pain, Stiffness, Function; Joint Pain; Hot Flashes; Hot Flash; Night Sweats; Vasomotor Symptoms
Keywords: Postmenopausal; Post menopause; Vasomotor Symptoms; Night sweats; Hot Flashes; Joint Pain; Joint Discomfort; Non-hormonal Treatment; Supplement
MeSH Terms: conditions — Arthralgia; Hot Flashes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JDS-HF3.0 Active Group (Active Comparator): Group of participants supplementing with JDS-HF3.0
  Interventions: Dietary Supplement: JDS-HF3.0
- Placebo Comparator (Placebo Comparator): Group consuming nonactive placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: JDS-HF3.0 — Active Supplement JDS-HF3.0
  Arms: JDS-HF3.0 Active Group
Other: Placebo — Nonactive Placebo
  Arms: Placebo Comparator

SUMMARY:
The goal of this interventional study is to evaluate whether the study product can help improve quality of life and reduce common menopause symptoms-such as joint discomfort, hot flashes and night sweats-in women aged 50-70. The primary research question is whether taking the study product daily for 12 weeks can reduce the severity and frequency of menopause-related symptoms.

DETAILED DESCRIPTION:
About 250 women across the U.S. will take part in this study. Participants will be randomly placed into one of two groups-one will take the active study product, and the other will take a placebo. All participants will take two tablets each morning for about 12 weeks. The total time the participant will be in the study is about 14 weeks, including the time it takes to collect baseline values.

All parts of the study are done virtually, in-person visits are not required. The participant will take part in five virtual check-ins, including a screening visit, a baseline visit, two check-ins during the study, and a final visit at the end. Throughout the study, the participant will be asked to complete daily diaries and weekly and monthly questionnaires to report on their symptoms and how they are feeling. These will include questions about hot flashes, night sweats, physical comfort, and overall well-being. The study is led by a research team based in Harrison, NY, USA.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy biological females who are 50-70 years of age (inclusive).
2. Have a body mass index (BMI) between 18.5 to 34.9 kg/m2 (inclusive).
3. Self-reported as postmenopause. Defined as 12 months without a menstrual cycle in individuals who undergo "Natural" Menopause (Not Surgically or medically induced) and who have self-reported menopausal outcomes for the past 6 months.
4. Have self-reported menopause related joint outcomes of moderate or severe severity according to a perceived discomfort greater or equal to 5 and less than 10 on a scale of 0-10 (participants rating their discomfort 5-9 will be included).
5. Have self-reported > or equal to 4 hot flashes on average per day.
6. In good general health (no active or uncontrolled diseases or conditions) and able to consume the study product.
7. Agree to refrain from treatments listed in Section 6.5 in the defined timeframe.
8. Have reliable, stable access to Wi-Fi and a smart phone/device.
9. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

1. Individuals who are lactating, pregnant, or planning to become pregnant during the study.
2. Active participation in a clinical trial.
3. Use of any treatment for menopausal outcomes or other concomitant treatments for menopausal symptoms, joint health or at the discretion of the investigator. (Participants may be deemed ineligible at the discretion of the investigator if the medication may cause adverse interaction.)
4. Have a known sensitivity, intolerability, or allergy to any of the study product or their excipients.
5. Use of Glucosamine and/or Chondroitin for joint outcomes in the last 3 months prior to screening.
6. Received a COVID-19 vaccine in the 2 weeks prior to screening or during the study period, current COVID-19 infections or currently have the post-COVID-19 condition as defined by World Health Organization (WHO) (i.e., individuals with a history of probable or confirmed SARS-CoV-2 infection, usually 3 months from the onset of COVID-19 with symptoms that last for at least two months and cannot be explained by an alternative diagnosis).
7. Have a positive medical history of heart disease, renal disease, hepatic impairment, or active systemic infection (i.e., Lyme disease, TB, HIV).
8. History of cancer (except localized skin cancer without metastases) within two (2) years prior to screening.
9. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential subject at risk because of participation in the study or influence the results or the potential subject's ability to participate in the study.
10. History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs (i.e., Crohn's disease, short bowel, acute or chronic pancreatitis, gastric bypass procedures, or pancreatic insufficiency).
11. Participant has an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea).
12. Major surgery in three months prior to screening or planned major surgery during the study.
13. History of alcohol or substance abuse in the last 5 years.
14. Has evidence of inflammatory rheumatic disease or other diagnosed anti-inflammatory disease.
15. Has evidence of autoimmune disease(s).
16. Chronic use of curcumin or curcuminoids in an herbal or dietary supplement. Note: Screened participants that are willing to undergo a washout period of at least 3 months prior to participation in the trial can be enrolled.
17. Chronic pain medication and use of analgesics specifically for joint-related discomfort (i.e. Opiates, Tramadol) Note: Screened participants that are willing to undergo a washout period of at least 2 weeks during the duration of the trial can be enrolled.
18. Have severe joint and/or severe bone deformities.
19. Diagnosed bone fractures.
20. Are a candidate for surgical joint replacement.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender Female
Enrollment: 250 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Menopause Related Quality of Life Outcomes | From enrollment to the end of study at 12 weeks
  Change from baseline in scores for severity of perceived joint discomfort, frequency of perceived joint discomfort, perceived joint mobility and perceived daily mobility assessed via a Visual Analog Scale (VAS). Response options will range from 0-100, with a higher score reflecting the worse outcome.
Change from Baseline in Menopause Related Quality of Life Outcomes | From enrollment to the end of study at 12 weeks
  Change from baseline in scores for Arthralgia Inventory (PRAI) score. The rating scale ranges from 0-10, with a higher score indicating a worse outcome.
Change from Baseline in Menopause Related Quality of Life Outcomes | From enrollment to the end of study at 12 weeks
  Change from baseline in scores for Musculoskeletal Health Questionnaire (MSK-HQ) score. Each response ranges from "not at all" to "very severe", with a higher score indicating a better outcome.

SECONDARY OUTCOMES:
Change from Baseline on Overall Menopausal Symptoms | From enrollment to the end of study at 12 weeks
  Change from baseline in scores for the following: Menopause Specific Quality of Life Questionnaire (MENQOL). Each question being scored from 0 to 6, with 6 being the worse outcome.
Change from Baseline on Overall Menopausal Symptoms | From enrollment to the end of study at 12 weeks
  Change from baseline in scores for Menopausal Rating Scale (MRS).Each question is rated on a 5-point scale with the higher number correlating with the more severe symptoms and worse outcome.
Change from Baseline on Overall Menopausal Symptoms | From enrollment to the end of study at 12 weeks
  Change from baseline in the frequency of menopause related hot flashes assessed via daily diaries. Daily diaries include the number of total vasomotor occurrences, the severity of total vasomotor occurrences and the number of times awoke during the night due to night sweat occurrences.

OTHER OUTCOMES:
Reports of Adverse Events | From baseline to the end of study at 12 weeks
  Assess the safety and tolerability of the study product in healthy participants

CONTACTS AND LOCATIONS:
Locations (1):
- Bonafide Health, Harrison, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will be privately owned.

REFERENCES:
- [Background] Heinemann K, Ruebig A, Potthoff P, Schneider HP, Strelow F, Heinemann LA, Do MT. The Menopause Rating Scale (MRS) scale: a methodological review. Health Qual Life Outcomes. 2004 Sep 2;2:45. doi: 10.1186/1477-7525-2-45. PMID 15345062
- [Background] Shep D, Khanwelkar C, Gade P, Karad S. Efficacy and safety of combination of curcuminoid complex and diclofenac versus diclofenac in knee osteoarthritis: A randomized trial. Medicine (Baltimore). 2020 Apr;99(16):e19723. doi: 10.1097/MD.0000000000019723. PMID 32311961
- [Background] Shep D, Khanwelkar C, Gade P, Karad S. Safety and efficacy of curcumin versus diclofenac in knee osteoarthritis: a randomized open-label parallel-arm study. Trials. 2019 Apr 11;20(1):214. doi: 10.1186/s13063-019-3327-2. PMID 30975196
- [Background] Kumar N, Singh S, Patro N, Patro I. Evaluation of protective efficacy of Spirulina platensis against collagen-induced arthritis in rats. Inflammopharmacology. 2009 Jun;17(3):181-90. doi: 10.1007/s10787-009-0004-1. Epub 2009 Apr 24. PMID 19390977
- [Background] Dillon JC, Phuc AP, Dubacq JP. Nutritional value of the alga Spirulina. World Rev Nutr Diet. 1995;77:32-46. doi: 10.1159/000424464. No abstract available. PMID 7732699
- [Background] Castel LD, Wallston KA, Saville BR, Alvarez JR, Shields BD, Feurer ID, Cella D. Validity and reliability of the Patient-Reported Arthralgia Inventory: validation of a newly-developed survey instrument to measure arthralgia. Patient Relat Outcome Meas. 2015 Jul 28;6:205-14. doi: 10.2147/PROM.S47997. eCollection 2015. PMID 26251635
- [Background] Magni A, Agostoni P, Bonezzi C, Massazza G, Mene P, Savarino V, Fornasari D. Management of Osteoarthritis: Expert Opinion on NSAIDs. Pain Ther. 2021 Dec;10(2):783-808. doi: 10.1007/s40122-021-00260-1. Epub 2021 Apr 19. PMID 33876393
- [Background] Suhail M, Rehan M, Tarique M, Tabrez S, Husain A, Zughaibi TA. Targeting a transcription factor NF-kappaB by green tea catechins using in silico and in vitro studies in pancreatic cancer. Front Nutr. 2023 Jan 11;9:1078642. doi: 10.3389/fnut.2022.1078642. eCollection 2022. PMID 36712528
- [Background] Ahmed S. Green tea polyphenol epigallocatechin 3-gallate in arthritis: progress and promise. Arthritis Res Ther. 2010;12(2):208. doi: 10.1186/ar2982. Epub 2010 Apr 28. PMID 20447316
- [Background] Zaratin P, Angelici O, Clarke GD, Schmid G, Raiteri M, Carita F, Bonanno G. NK3 receptor blockade prevents hyperalgesia and the associated spinal cord substance P release in monoarthritic rats. Neuropharmacology. 2000;39(1):141-9. doi: 10.1016/s0028-3908(99)00087-8. PMID 10665827
- [Background] Barbalho S. M., Goulart R. D. A, Buglio D. S., Araujo A. C., Guiguer E. L. The possible role of green tea on osteoarthritis: a narrative report. Longhua Chin Med 2020;3:11.
- [Background] Strand NH, D'Souza RS, Gomez DA, Whitney MA, Attanti S, Anderson MA, Moeschler SM, Chadwick AL, Maloney JA. Pain during menopause. Maturitas. 2025 Jan;191:108135. doi: 10.1016/j.maturitas.2024.108135. Epub 2024 Oct 31. PMID 39500125
- [Background] Magliano M. Menopausal arthralgia: Fact or fiction. Maturitas. 2010 Sep;67(1):29-33. doi: 10.1016/j.maturitas.2010.04.009. PMID 20537472
- [Background] Blumer J. Arthralgia of menopause - A retrospective review. Post Reprod Health. 2023 Jun;29(2):95-97. doi: 10.1177/20533691231172565. Epub 2023 May 1. PMID 37127408
- See also: Epigallocatechin-3-gallate (EGCG): Chemical and biomedical perspectives — https://doi.org/10.1016/j.phytochem.2006.06.020
- See also: Corticosteroid Adverse Effects — https://www.ncbi.nlm.nih.gov/books/NBK531462/
- See also: Green tea polyphenol epigallocatechin 3-gallate in arthritis: progress and promise. — https://doi.org/10.1186/ar2982
- See also: Measurement properties of the musculoskeletal health questionnaire (MSK-HQ): a between country comparison — https://pubmed.ncbi.nlm.nih.gov/32576190/
- See also: The potential application of Spirulina (Arthrospora) as a nutritional and therapeutic supplement in health management — https://www.algbiotek.com/bilimsel/PDF%20Dosyalarrrrrr/sagliktaspirulinaninbesinselveterapotiktakviyeolarakpotansiyelkullanimi.pdf